CLINICAL TRIAL: NCT02327390
Title: Phase I Study Using Autologous Ex Vivo-Activated (X-ACT) Lymph Node Lymphocytes as Adoptive Immunotherapy in Advanced Malignant Melanoma Patients
Brief Title: Ex Vivo-Activated Lymph Node Lymphocytes in Treating Patients With Stage IIIC-IV Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Left
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3612; NCI-2014-00761 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 3612 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-12-17; First posted 2014-12-30 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Stage IIIC Skin Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- X-ACT lymph node cell dose and schedule (Experimental): All patients will begin at dose level 1 and will be moved to higher dosing levels as long as the patient does not experience two or more dose limiting toxicities and maintains an acceptable performance status. A minimum of three patients will be enrolled per dose level and no patients will be enrolled on higher dose levels if dose limiting toxicities are encountered.
  Dose level 1: 0.5 x 10^10 X-ACT cells. 2 infusions 4 weeks apart
  Dose level 2: 1.0 x 10^10 X-ACT cells. 1 infusion
  Dose level 3: 0.5 x 10^10 X-ACT cells. 4 infusions 4 weeks apart
  Dose level 4: 1.0 x 10^10 X-ACT cells. 2 infusions 4 weeks apart
  Dose level -1: 0.5 x 10^10 X-ACT cells. 1 infusion (if necessary)
  Interventions: Procedure: lymph node; Biological: X-ACT

INTERVENTIONS:
Procedure: lymph node — Undergo surgery to remove a melanoma-draining lymph node for generation of X-ACT cells in the laboratory
  Other Names: lymph node excisional biopsy
Biological: X-ACT — Administered as an IV infusion
  Other Names: ex vivo-activated autologous lymph node lymphocytes; X-ACT autologous lymph node lymphocytes

SUMMARY:
This phase I trial studies the safety and best dose of ex-vivo activated lymph node lymphocytes (X-ACT) as well as how well the immune system responds to X-ACT treatment in participants with stage IIIC-IV melanoma. X-ACT treatment involves removing a participant's lymph node(s) close to a melanoma tumor. These lymph nodes contain special kind of cells (called T cells) which can be activated (getting the cells to start up certain responses in the immune system) outside of the body in an approved laboratory. The activated T cells are then injected back into the same participant using an i.v. to help the participant's immune system to target melanoma. The participant will undergo regular blood testing to determine whether the X-ACT treatment has resulted in changes to the immune system and also whether the T cells which were given back to the patient persist in the blood stream over time. In addition, the effect of the X-ACT treatment on the growth or shrinkage of the participant's melanoma will be measured.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and toxicity profile of repeated infusions of ex-vivo activated tumor-draining lymphocytes (X-ACT) in participants with advanced melanoma.

SECONDARY OBJECTIVES:

I. Assess the feasibility of multiple infusions of X-ACT. II. Assess the effect of dose and schedule on immunologic parameters using two novel biomarkers.

III. Observe the clinical outcomes of participants receiving X-ACT therapy.

OUTLINE: This is a dose-escalation study.

STEP 1: Participants undergo lymph node biopsy for collection of at least one melanoma-draining lymph node (MDLN). MDLN cells will then be cryopreserved into aliquots until they are needed to generate an activated T cell culture.

STEP 2: Cryopreserved lymph node cells are thawed and then undergo activation with anti-cluster of differentiation (CD)3/anti-CD28 microbeads. The cultures then undergo expansion over 14-18 days in the presence of recombinant human interleukin-2 and anti-vascular endothelial growth factor antibody. The activated X-ACT cells are then transferred i.v. into the same participant from which they were derived with no additional therapy.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1

  * Participants must have a histologic diagnosis of melanoma either from a primary or metastatic site; Participants with brain metastases must have completed radiation therapy >30 days prior to enrollment
  * Participants must have American Joint Committee on Cancer (AJCC) stage IIIC unresected or IV disease
  * Patients with non-measureable or measurable disease are eligible. Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter for non-nodal lesions and short axis for nodal lesions to be recorded) as ≥ 20 mm by chest x-ray, as ≥ 10 mm with CT scan, or ≥ 10 mm with calipers by clinical exam. Malignant lymph nodes, to be considered pathologically enlarged and measurable, must be ≥ 15 mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

    * Tumor lesions that are situated in a previously irradiated area can be considered measurable as long as ≥ 30 days has passed since radiation to that area
  * Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
  * Life expectancy (untreated) of > 4 months, in the opinion of and as documented by the investigator
  * White blood count > 3,000/mcL
  * Absolute neutrophil count > 1,200/mcL
  * Platelet count > 100,000/mcL
  * Serum creatinine < 2.0 mg/dL
  * International normalized ratio (INR) ≤ 2.0
  * In the opinion of the investigator, participant must be medically fit to undergo surgical procedure
  * Participants treated with prior chemotherapy, cytotoxic chemotherapy, radiation, biotherapy, or any investigational agent > 30 days prior to lymph node removal are eligible
  * Women of child-bearing potential must agree to use adequate contraception (double barrier method of birth control or abstinence) during participation in the study; should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately
  * Participants must be disease free of prior invasive malignancies for > 5 years, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or cancer in-situ of the cervix
  * Participants must be able to understand and willing to sign a written informed consent document
* STEP 2

  * Successful removal of melanoma-draining lymph node (MDLN)
  * ECOG Performance status ≤ 1
  * White blood count > 3,000/mcL
  * Absolute neutrophil count > 1,500/mcL
  * Platelet count > 100,000/mcL
  * Serum creatinine < 2.0 mg/dL
  * Serum direct bilirubin < 2 x institutional upper limit of normal
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])
  * Alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal
  * Participants with liver metastases who do not meet the eligibility parameters may only be enrolled at the discretion of the principal investigator (PI)

Exclusion Criteria:

Step 1

* Participants who are taking immunosuppressive medications that cannot be discontinued (corticosteroids); participants who have discontinued immunosuppressive medications but be at least 1 week post their last dose. Patients who are taking physiologic replacement doses of corticosteroids equivalent to oral prednisone 10 mg per day will not be excluded.
* Participants who are receiving any other investigational agents
* Participants with a history of autoimmune disease requiring continuous treatment
* Participants receiving any medications or substances to treat active infection
* Pregnant or breastfeeding
* Participants with human immunodeficiency virus (HIV) or hepatitis, or known active cytomegalovirus (CMV), Epstein-Barr virus (EBV) or any other viral illness requiring treatment are ineligible because of the potential for pharmacokinetic interactions with ACT lymph node lymphocytes
* Any condition or behavior that in the judgment of the investigator, would compromise the participant's ability to participate in the study and/or comply with study procedures
* Patients with bleeding disorders are ineligible due to lymph node removal possibly causing excessive bleeding. Bleeding disorder will be defined by an INR level of > 2.0

Step 2 None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2016-07-18 (Actual); Study Completion 2016-07-18 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | At least 30 days after last infusion
  Number of patients with dose-limiting toxicity will be reported for each treatment group. Maximum tolerated dose may be determined if dose-limiting toxicity is observed.

SECONDARY OUTCOMES:
Prevalence of each biomarker in peripheral blood over time | Up to 1 year
  The temporal profiles of the two biomarkers will be summarized as mean +/- standard deviation at each time point and visualized using scatter plot stratified by dose level and schedule.
Clinical response defined by Response Evaluation Criteria In Solid Tumors 1.1 | Up to 1 year
  Will be estimated based on the number of clinical responses observed using a binomial distribution and its confidence intervals will be estimated using Wilson's method. A complete response (CR) is defined as the disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10mm. A partial response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. Stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Kim, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States